CLINICAL TRIAL: NCT07167056
Title: Artificial Intelligence-Powered Support For Quality Of Life Improvement In Patients With Cancer
Brief Title: Artificial Intelligence-Powered Support For Quality Of Life Improvement In Participants With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Florida Department of Health (Casey DeSantis Florida Cancer Innovation Fund) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE10Z25
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Psychotherapy; Mental health; Distress; Stage I Cancer; Stage II Cancer; Stage III Cancer; Chatbot; Artificial Intelligence; AI
MeSH Terms: conditions — Neoplasms; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychotherapy + WYSA App (Experimental)
  Interventions: Behavioral: Standard of Care Psychotherapy; Behavioral: WYSA App
- Standard of Care Psychotherapy (Active Comparator)
  Interventions: Behavioral: Standard of Care Psychotherapy

INTERVENTIONS:
Behavioral: Standard of Care Psychotherapy — Participants will receive six psychotherapy sessions over the course of approximately 3 months.
Behavioral: WYSA App — Participants will have access to the WYSA mental health support artificial intelligence app over the course of the 3 months that they are participating in psychotherapy sessions per standard of care. The app will contain features intended to manage symptoms of depression and anxiety in individuals with cancer. The app will include an AI-powered chatbot with Cognitive Behavioral Therapy (CBT) and mindfulness techniques, visual progress elements (a progress roadmap, a weekly progress report, etc.), and a customizable tool library. Participants are instructed to use the app whenever they feel like it, if they are in distress, or if the app prompts them to use it. App prompts (notifications) will occur once daily.
  Arms: Psychotherapy + WYSA App

SUMMARY:
This research study is for people who are diagnosed with cancer and are receiving treatment for cancer who may benefit from psychotherapy. The purpose of the study is to see whether an artificial intelligence (AI) powered application (app) could help improve quality of life, anxiety symptoms, and/or depression symptoms, over the course of psychotherapy sessions. Participants in this study will be randomly assigned to one of two groups. One group will receive psychotherapy per usual care and will receive access to the AI-powered app. The second group will only receive psychotherapy per usual care and will NOT receive access to the AI-powered app. Both groups will complete surveys about their quality of life, anxiety symptoms, and depression symptoms over the course of their psychotherapy visits.

DETAILED DESCRIPTION:
Getting a cancer diagnoses and going through treatment can be difficult and lead to symptoms of distress, like anxiety and depression. Feeling distressed or upset can make people with cancer feel worse and potentially shorten how long they live. Because of this, it is important to address the distress that people with cancer may feel in order to improve their well-being. Treatments that don't use medication, like psychotherapy ("talk therapy), relaxation techniques, and mindfulness, can help reduce distress in people with cancer. However, some people do not have access to these types of things, and mental health care overall can be limited by financial, logistical, and geographical barriers. One solution to these barriers could be artificial intelligence (AI)-powered interventions using mobile applications (apps) on someone's phone. AI tools, like chatbots, can provide personal support. They can use Cognitive Behavioral Therapy (CBT) and mindfulness to provide support. They can also provide tools to track someone's mood. AI tools do not replace a diagnosis from a doctor or treatment from a doctor or other clinical care provider. However, these tools could still support and help to improve someone's mental health and well-being. People who have studied this have found that this day-to-day support has decreased anxiety and depression in the general population. However, the use of AI tools to support mental health in people with cancer is not yet well studied.

WYSA is an AI-powered chatbot that uses evidence-based techniques like Cognitive Behavioral Therapy (CBT) and mindfulness. For the purposes of this study, WYSA will be used in addition to standard of care psychotherapy. WYSA will not replace psychotherapy care in this study, and it will not replace a doctor's advice or diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Participants in active cancer treatment (receiving chemotherapy, immunotherapy and/or radiation therapy) AND reporting National Comprehensive Cancer Network (NCCN) Distress Thermometer scores ≥4. The NCCN Distress Thermometer is a validated, single-item screening tool routinely used in cancer care at Cleveland Clinic Florida to identify individuals experiencing psychological distress. A score of 4 or higher indicates clinically significant distress and serves as the eligibility threshold for enrollment in this study.
* Participants followed by a medical oncologist, radiation oncologist, and/or surgical oncologist of any subspecialty at Cleveland Clinic Florida and have no barrier to receive psychotherapy care (e.g. no insurance restrictions)
* Participants with biopsy proven cancer of any type, stages I-III.
* Adults aged 18 years or older.
* Able to understand and read English and/or Spanish.
* Participants who own a smartphone compatible with the mobile app (Android or IOS) or have regular (Daily) access to one.
* Participants who are willing and able to provide informed consent.

Exclusion Criteria:

* Age <18 years.
* Participants with stage 4 cancer.
* Participants with active severe psychiatric conditions identified by the Cleveland Clinic psychotherapist as any diagnoses that could significantly impair a participant's ability to engage meaningfully with the intervention or provide informed consent. These include, but are not limited to:

  * Current or recent (within the past 6 months) psychotic disorders (e.g., schizophrenia, schizoaffective disorder)
  * Bipolar disorder in a manic or severe depressive phase
  * Active suicidal ideation with intent or recent suicide attempt (within the past 6 months)
  * Severe cognitive impairment or neurocognitive disorders that compromise comprehension or communication or interferes with chatbot use.
  * Any condition requiring psychiatric hospitalization within the past 6 months
* Concurrent enrollment in another trial targeting psychological distress to avoid bias.
* Limited life expectancy (<3 months) as determined by the oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.

SECONDARY OUTCOMES:
Change in Anxiety | Baseline, 3 months
  Anxiety is measured by the Generalized Anxiety Disorder-7 (GAD-7) questionnaire. The questionnaire contains 7 questions asking participants about their anxiety symptoms on a 4-point Likert scale from "Not at all" (0) to "Nearly every day" (3). There is one questions regarding how difficult these symptoms have made daily life, where participants provide an answer on a 4-point scale from "Not difficult at all" to "Extremely difficult." Higher scores indicate greater anxiety symptoms.
Change in Depression | Baseline, 3 months
  Depression is measured by the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 contains 8 questions asking participants about their depression symptoms on a 4-point Likert scale from "Not at all" (0) to "Nearly every day" (3). There is one questions regarding how difficult these symptoms have made daily life, where participants provide an answer on a 4-point scale from "Not difficult at all" to "Extremely difficult." Higher scores indicate greater depression symptoms.
Change in physical functioning | Baseline, 3 months
  Physical functioning is measured by the physical functioning (functional scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains five questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate lower physical functioning.
Change in role functioning | Baseline, 3 months
  Role functioning is measured by the role functioning (functional scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains two questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate lower role functioning.
Change in emotional functioning | Baseline, 3 months
  Emotional functioning is measured by the emotional functioning (functional scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains four questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate lower emotional functioning.
Change in cognitive functioning | Baseline, 3 months
  Cognitive functioning is measured by the cognitive functioning (functional scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains two questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate lower cognitive functioning.
Change in social functioning | Baseline, 3 months
  Social functioning is measured by the social functioning (functional scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains two questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate lower social functioning.
Change in fatigue | Baseline, 3 months
  Fatigue is measured by the fatigue (symptom scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains three questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater fatigue symptoms.
Change in nausea/vomiting | Baseline, 3 months
  Nausea/vomiting is measured by the nausea and vomiting (symptom scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains two questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater fatigue symptoms.
Change in pain | Baseline, 3 months
  Pain is measured by the pain (symptom scale) subscale of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It contains two questions, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater fatigue symptoms.
Change in dyspnea | Baseline, 3 months
  Dyspnea is measured by the dyspnea (symptom item) item of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It is one question, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater dyspnea symptoms.
Change in insomnia | Baseline, 3 months
  Insomnia is measured by the insomnia (symptom item) item of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It is one question, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater insomnia symptoms.
Change in appetite loss | Baseline, 3 months
  Appetite loss is measured by the appetite loss (symptom item) item of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It is one question, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater appetite loss symptoms.
Change in constipation | Baseline, 3 months
  Constipation is measured by the constipation (symptom item) item of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It is one question, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater constipation symptoms.
Change in diarrhea | Baseline, 3 months
  Diarrhea is measured by the diarrhea (symptom item) item of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It is one question, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater diarrhea symptoms.
Change in financial difficulties | Baseline, 3 months
  Financial difficulties is measured by the financial difficulties (symptom item) item of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 questionnaire. It is one question, where participants provide an answer on a 4-point Likert scale from "Not at all" (1) to "Very Much" (4). Higher scores indicate greater financial difficulties.
Engagement, measured by frequency of use of app | Length of participation, up to 3 months
  Frequency will be measured by the amount of times that participants use the app, recorded as the date/time of usage
Engagement, measured by tool usage in app | Length of participation, up to 3 months
  The app contains tools related to mindfulness and Cognitive Behavioral Therapy (CBT)-informed approaches. Engagement is measured by frequency of tool usage.
Engagement, measured by length of app chatbot interaction | Length of participation, up to 3 months
  "Length" is defined as number of messages exchanged during chatbot interaction.
Incidence of adverse events (AEs) | One month after completion of participation, up to 4 months
Change in Quality of Life, according to number of psychotherapy visits completed | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of gender | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of race | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of ethnicity | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of marital status | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of cancer type | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of cancer stage | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of time since diagnosis | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of comorbidities | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of insurance status | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of in-person vs virtual psychotherapy visit | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of current therapy regimen | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of current psychiatric medication | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of current mental health diagnosis | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.
Change in Quality of Life, according to participant characteristic of number of psycho-oncology visits attended previously | Baseline, 3 months
  Quality of life (QoL) is measured by the global health status/QoL subscale of the EORTC QLQ-C30 version 3.0 questionnaire. The global health status/QoL subscale contains two questions, where participants provide an answer on a 7-point Likert scale from "Very poor" (1) to "Excellent" (7). Higher scores indicate greater global health status/QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD, FACP, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson LE, Waller A, Mitchell AJ. Screening for distress and unmet needs in patients with cancer: review and recommendations. J Clin Oncol. 2012 Apr 10;30(11):1160-77. doi: 10.1200/JCO.2011.39.5509. Epub 2012 Mar 12. PMID 22412146
- [Background] Kroenke K, Theobald D, Wu J, Loza JK, Carpenter JS, Tu W. The association of depression and pain with health-related quality of life, disability, and health care use in cancer patients. J Pain Symptom Manage. 2010 Sep;40(3):327-41. doi: 10.1016/j.jpainsymman.2009.12.023. Epub 2010 Jun 26. PMID 20580201
- [Background] Niedzwiedz CL, Knifton L, Robb KA, Katikireddi SV, Smith DJ. Depression and anxiety among people living with and beyond cancer: a growing clinical and research priority. BMC Cancer. 2019 Oct 11;19(1):943. doi: 10.1186/s12885-019-6181-4. PMID 31604468
- [Background] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- [Background] Brown KW, Levy AR, Rosberger Z, Edgar L. Psychological distress and cancer survival: a follow-up 10 years after diagnosis. Psychosom Med. 2003 Jul-Aug;65(4):636-43. doi: 10.1097/01.psy.0000077503.96903.a6. PMID 12883115
- [Background] Gao W, Bennett MI, Stark D, Murray S, Higginson IJ. Psychological distress in cancer from survivorship to end of life care: prevalence, associated factors and clinical implications. Eur J Cancer. 2010 Jul;46(11):2036-44. doi: 10.1016/j.ejca.2010.03.033. Epub 2010 May 4. PMID 20447824
- [Background] Phoosuwan N, Lundberg PC. Psychological distress and health-related quality of life among women with breast cancer: a descriptive cross-sectional study. Support Care Cancer. 2022 Apr;30(4):3177-3186. doi: 10.1007/s00520-021-06763-z. Epub 2021 Dec 23. PMID 34950961
- [Background] Pinquart M, Duberstein PR. Depression and cancer mortality: a meta-analysis. Psychol Med. 2010 Nov;40(11):1797-810. doi: 10.1017/S0033291709992285. Epub 2010 Jan 20. PMID 20085667
- [Background] Satin JR, Linden W, Phillips MJ. Depression as a predictor of disease progression and mortality in cancer patients: a meta-analysis. Cancer. 2009 Nov 15;115(22):5349-61. doi: 10.1002/cncr.24561. PMID 19753617
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Kubo A, Kurtovich E, McGinnis M, Aghaee S, Altschuler A, Quesenberry C Jr, Kolevska T, Avins AL. A Randomized Controlled Trial of mHealth Mindfulness Intervention for Cancer Patients and Informal Cancer Caregivers: A Feasibility Study Within an Integrated Health Care Delivery System. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419850634. doi: 10.1177/1534735419850634. PMID 31092044
- [Background] Lei Chui P, Wai S, Lai LL, See MH, Tan SB. Mindful Breathing: Effects of a Five-Minute Practice on Perceived Stress and Mindfulness Among Patients With Cancer. Clin J Oncol Nurs. 2021 Apr 1;25(2):174-180. doi: 10.1188/21.CJON.174-180. PMID 33739333
- [Background] Ngamkham S, Holden JE, Smith EL. A Systematic Review: Mindfulness Intervention for Cancer-Related Pain. Asia Pac J Oncol Nurs. 2019 Apr-Jun;6(2):161-169. doi: 10.4103/apjon.apjon_67_18. PMID 30931361
- [Background] Biddell CB, Waters AR, Angove RSM, Gallagher KD, Rosenstein DL, Spees LP, Kent EE, Planey AM, Wheeler SB. Facing financial barriers to healthcare: patient-informed adaptation of a conceptual framework for adults with a history of cancer. Front Psychol. 2023 May 15;14:1178517. doi: 10.3389/fpsyg.2023.1178517. eCollection 2023. PMID 37255517
- [Background] Faller H, Schuler M, Richard M, Heckl U, Weis J, Kuffner R. Effects of psycho-oncologic interventions on emotional distress and quality of life in adult patients with cancer: systematic review and meta-analysis. J Clin Oncol. 2013 Feb 20;31(6):782-93. doi: 10.1200/JCO.2011.40.8922. Epub 2013 Jan 14. PMID 23319686
- [Background] Smith SK, Nicolla J, Zafar SY. Bridging the gap between financial distress and available resources for patients with cancer: a qualitative study. J Oncol Pract. 2014 Sep;10(5):e368-72. doi: 10.1200/JOP.2013.001342. Epub 2014 May 27. PMID 24865219
- [Background] Chang CL, Sinha C, Roy M, Wong JCM. AI-Led Mental Health Support (Wysa) for Health Care Workers During COVID-19: Service Evaluation. JMIR Form Res. 2024 Apr 19;8:e51858. doi: 10.2196/51858. PMID 38640476
- [Background] Durden E, Pirner MC, Rapoport SJ, Williams A, Robinson A, Forman-Hoffman VL. Changes in stress, burnout, and resilience associated with an 8-week intervention with relational agent "Woebot". Internet Interv. 2023 Jun 14;33:100637. doi: 10.1016/j.invent.2023.100637. eCollection 2023 Sep. PMID 37635948
- [Background] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005
- [Background] Inkster B, Sarda S, Subramanian V. An Empathy-Driven, Conversational Artificial Intelligence Agent (Wysa) for Digital Mental Well-Being: Real-World Data Evaluation Mixed-Methods Study. JMIR Mhealth Uhealth. 2018 Nov 23;6(11):e12106. doi: 10.2196/12106. PMID 30470676
- [Background] Leo AJ, Schuelke MJ, Hunt DM, Metzler JP, Miller JP, Arean PA, Armbrecht MA, Cheng AL. A Digital Mental Health Intervention in an Orthopedic Setting for Patients With Symptoms of Depression and/or Anxiety: Feasibility Prospective Cohort Study. JMIR Form Res. 2022 Feb 21;6(2):e34889. doi: 10.2196/34889. PMID 35039278
- [Background] Leo AJ, Schuelke MJ, Hunt DM, Miller JP, Arean PA, Cheng AL. Digital Mental Health Intervention Plus Usual Care Compared With Usual Care Only and Usual Care Plus In-Person Psychological Counseling for Orthopedic Patients With Symptoms of Depression or Anxiety: Cohort Study. JMIR Form Res. 2022 May 4;6(5):e36203. doi: 10.2196/36203. PMID 35507387
- [Background] Cheng AL, Leo AJ, Calfee RP, Dy CJ, Armbrecht MA, Abraham J. Multi-stakeholder perspectives regarding preferred modalities for mental health intervention delivered in the orthopedic clinic: a qualitative analysis. BMC Psychiatry. 2023 May 19;23(1):347. doi: 10.1186/s12888-023-04868-9. PMID 37208668
- [Background] Davis A, Landers SE, Sun Y, Nguyen VO, Bolger N, Lewis RA, Rosenthal SL. Evaluating the Feasibility and Acceptability of a Mobile Mental Health Intervention for Adolescent Depression and Anxiety. Clin Pediatr (Phila). 2026 Jan;65(1):53-62. doi: 10.1177/00099228251371903. Epub 2025 Sep 7. PMID 40914852
- [Background] Phang YS, Heaukulani C, Martanto W, Morris R, Tong MM, Ho R. Perceptions of a Digital Mental Health Platform Among Participants With Depressive Disorder, Anxiety Disorder, and Other Clinically Diagnosed Mental Disorders in Singapore: Usability and Acceptability Study. JMIR Hum Factors. 2023 Mar 29;10:e42167. doi: 10.2196/42167. PMID 36989020
- [Background] Dinesh DN, Rao MN, Sinha C. Language adaptations of mental health interventions: User interaction comparisons with an AI-enabled conversational agent (Wysa) in English and Spanish. Digit Health. 2024 May 24;10:20552076241255616. doi: 10.1177/20552076241255616. eCollection 2024 Jan-Dec. PMID 38798884
- [Background] Aghakhani S, Carre N, Mostovoy K, Shafer R, Baeza-Hernandez K, Entenberg G, Testerman A, Bunge EL. Qualitative analysis of mental health conversational agents messages about autism spectrum disorder: a call for action. Front Digit Health. 2023 Dec 5;5:1251016. doi: 10.3389/fdgth.2023.1251016. eCollection 2023. PMID 38116099
- [Background] Sinha C, Dinesh D, Heaukulani C, Phang YS. Examining a brief web and longitudinal app-based intervention [Wysa] for mental health support in Singapore during the COVID-19 pandemic: mixed-methods retrospective observational study. Front Digit Health. 2024 Dec 23;6:1443598. doi: 10.3389/fdgth.2024.1443598. eCollection 2024. PMID 39764209
- [Background] Aghakhani S, Rousseau A, Mizrahi S et al. Conversational Agent Utilization Patterns of Individuals with Autism Spectrum Disorder. Journal of Technology in Behavioral Science 2024.
- [Background] Iglesias M, Sinha C, Vempati R, Grace SE, Roy M, Chapman WC, Rinaldi ML. Evaluating a Digital Mental Health Intervention (Wysa) for Workers' Compensation Claimants: Pilot Feasibility Study. J Occup Environ Med. 2023 Feb 1;65(2):e93-e99. doi: 10.1097/JOM.0000000000002762. Epub 2022 Dec 2. PMID 36459701
- [Background] Beatty C, Malik T, Meheli S, Sinha C. Evaluating the Therapeutic Alliance With a Free-Text CBT Conversational Agent (Wysa): A Mixed-Methods Study. Front Digit Health. 2022 Apr 11;4:847991. doi: 10.3389/fdgth.2022.847991. eCollection 2022. PMID 35480848
- [Background] Malik T, Ambrose AJ, Sinha C. Evaluating User Feedback for an Artificial Intelligence-Enabled, Cognitive Behavioral Therapy-Based Mental Health App (Wysa): Qualitative Thematic Analysis. JMIR Hum Factors. 2022 Apr 12;9(2):e35668. doi: 10.2196/35668. PMID 35249886
- [Background] Meheli S, Sinha C, Kadaba M. Understanding People With Chronic Pain Who Use a Cognitive Behavioral Therapy-Based Artificial Intelligence Mental Health App (Wysa): Mixed Methods Retrospective Observational Study. JMIR Hum Factors. 2022 Apr 27;9(2):e35671. doi: 10.2196/35671. PMID 35314422
- [Background] Sinha C, Cheng AL, Kadaba M. Adherence and Engagement With a Cognitive Behavioral Therapy-Based Conversational Agent (Wysa for Chronic Pain) Among Adults With Chronic Pain: Survival Analysis. JMIR Form Res. 2022 May 23;6(5):e37302. doi: 10.2196/37302. PMID 35526201
- [Background] Gupta M, Malik T, Sinha C. Delivery of a Mental Health Intervention for Chronic Pain Through an Artificial Intelligence-Enabled App (Wysa): Protocol for a Prospective Pilot Study. JMIR Res Protoc. 2022 Mar 31;11(3):e36910. doi: 10.2196/36910. PMID 35314423
- [Background] Inkster B, Kadaba M, Subramanian V. Understanding the impact of an AI-enabled conversational agent mobile app on users' mental health and wellbeing with a self-reported maternal event: a mixed method real-world data mHealth study. Front Glob Womens Health. 2023 Jun 2;4:1084302. doi: 10.3389/fgwh.2023.1084302. eCollection 2023. PMID 37332481
- [Background] Inkster B, O'Brien R, Selby E, Joshi S, Subramanian V, Kadaba M, Schroeder K, Godson S, Comley K, Vollmer SJ, Mateen BA. Digital Health Management During and Beyond the COVID-19 Pandemic: Opportunities, Barriers, and Recommendations. JMIR Ment Health. 2020 Jul 6;7(7):e19246. doi: 10.2196/19246. PMID 32484783
- [Background] Sinha C, Meheli S, Kadaba M. Understanding Digital Mental Health Needs and Usage With an Artificial Intelligence-Led Mental Health App (Wysa) During the COVID-19 Pandemic: Retrospective Analysis. JMIR Form Res. 2023 Jan 26;7:e41913. doi: 10.2196/41913. PMID 36540052
- [Background] Kuchlous S, Kadaba M. Short Text Intent Classification for Conversational Agents. 2020 IEEE 17th India Council International Conference (INDICON). 2020:1-4.
- [Background] MacNeill AL, Doucet S, Luke A. Effectiveness of a Mental Health Chatbot for People With Chronic Diseases: Randomized Controlled Trial. JMIR Form Res. 2024 May 30;8:e50025. doi: 10.2196/50025. PMID 38814681
- [Background] Yoon S, Goh H, Low XC, Weng JH, Heaukulani C. User perceptions and utilisation of features of an AI-enabled workplace digital mental wellness platform 'mindline at work'. BMJ Health Care Inform. 2024 Aug 17;31(1):e101045. doi: 10.1136/bmjhci-2024-101045. PMID 39153756
- [Background] Weng JH, Hu Y, Heaukulani C, Tan C, Chang JK, Phang YS, Rajendram P, Tan WM, Loke WC, Morris RJT. Mental Wellness Self-Care in Singapore With mindline.sg: A Tutorial on the Development of a Digital Mental Health Platform for Behavior Change. J Med Internet Res. 2024 Jun 4;26:e44443. doi: 10.2196/44443. PMID 38833294